CLINICAL TRIAL: NCT06266598
Title: The Effect of Anti-diabetic Treatment Applied in Childhood Obesity on Zinc, Zinc α-2 Glycoprotein and Peroxisome Proliferation Activating Receptor-γ Levels
Brief Title: Effectiveness of Antidiabetic Treatment Applied in Childhood Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HÜMEYRA ACIKAN (Other)
Responsible Party: Sponsor-Investigator, HÜMEYRA ACIKAN, Research asistant, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-TF-HA-01
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Childhood Obesity; Insulin Resistance
Keywords: Obesity; Metformin; Biomarker
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Obesity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: In our study, there are 33 healthy children with normal weight (control group) and 52 obese children who will be treated with metformin. To observe the efficacy of the 3-month treatment before and after metformin treatment, Zn, Zinc α-2 Glycoprotein (ZAG), Peroxisome proliferation activating receptor γ (PPARγ), Leptin (LEP) and Adiponectin (ADIPO) levels were compared, as well as anthropometric measurements and routine biochemistry tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- obesity (Other): Children with obesity were recommended to have a diet appropriate for their age and gender and exercise at least 3 days a week for at least 60 minutes each time.
  All obese children under the age of 14 were started on metformin treatment at 1000 mg (500 mgx2) per day, and children over this age were started on metformin treatment at the adult dose of 2000 mg (1000 mgx2) per day.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Only obese children with insulin resistance were treated with metformin.

SUMMARY:
In our study, there are 33 healthy children with normal weight (control group) and 52 obese children who will be treated with metformin. To observe the efficacy of the 3-month treatment before and after metformin treatment, Zn, Zinc α-2 Glycoprotein (ZAG), Peroxisome proliferation activating receptor γ (PPARγ), Leptin (LEP) and Adiponectin (ADIPO) levels were compared, as well as anthropometric measurements and routine biochemistry tests.

ELIGIBILITY:
inclusion criteria:

* Body mass index (BMI) > 95th percentile
* Having insulin resistance
* Having a family history of Type 2 diabetes mellitus (T2DM)

exclusion criteria;

* Alcohol consumption and smoking
* Having T1DM and T2DM
* History of drug use

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-17 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (HOMA-IR) level | three months
  HOMA-IR is a condition in which the body's cells become less responsive to the effects of insulin. This means that the body needs more insulin to achieve the same effects, such as regulating blood sugar levels
Weight loss rate | three months
  Weight loss rate is typically defined as the amount of weight lost over a specific period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)